CLINICAL TRIAL: NCT03273504
Title: Efficacy Evaluation of the Activity of a Cosmetic Product (Topical Use) on Hair Regrowth vs Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1517
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hypertrichosis
MeSH Terms: conditions — Hypertrichosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actapil Corpo Spray (SHEDIR PHARMA Srl - Italy) (Experimental): Comparison within subjects of Actapil Corpo Spray versus Placebo. The study product will be applied twice a dayon the right or left leg (tibialis area) according to a randomisation list.
  The placebo product will be applied in the same way, on the controlateral leg.
  Interventions: Other: Actapil Corpo Spray (SHEDIR PHARMA Srl - Italy); Other: Placebo

INTERVENTIONS:
Other: Actapil Corpo Spray (SHEDIR PHARMA Srl - Italy) — The study product will be applied twice a day (at morning and at evening) for an interrupted period of 3 months, on the right or left leg (tibialis area) according to a randomisation list.
Other: Placebo — The placebo product will be applied twice a day (at morning and at evening) for an interrupted period of 3 months, on the controlateral leg (tibialis area) right or left leg according to a randomisation list.

SUMMARY:
Aim of the study is to evaluate clinically and by non-invasive instrumental evaluations the activity on hair regrowth of a topical cosmetic product versus placebo (comparison within subjects)

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* female sex
* with hypertrichosis
* agreeing not to perform epilation or scrub/peeling treatment on the test area (legs) during the week preceding the inclusion
* good general state of health

Exclusion Criteria:

* pregnancy
* lactation
* subjects whose insufficient adhesion to the study protocol is foreseeable
* sensitive skin
* oral contraceptive therapy started less than 1 year
* presence of varicose or capillary veins of surface
* hormonal therapies able to influence hair growth.
* presence of cutaneous disease on the tested area, as lesions, scars, malformations.
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* cancer.
* farmacological topical treatment and surgery and/or medical treatment on the treated side performed in the last 3 months
* systemic corticosteroids
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* diuretic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the hair density | Baseline (T0), 1 month (T1), 3 months (T3)
  Hair density (hair number/mm2) is calculate by Image-Pro Plus software on the microscopic images captured with Dino-Lite (AnMo Electronics Corporation,Taiwan)
Change from baseline of the percentage of terminal hair | Baseline (T0), 1 month (T1), 3 months (T3)
  Percentage of terminal hair (terminal hair has a diameter >0.04 mm) is calculate by Image-Pro Plus software on the microscopic images captured with Dino-Lite (AnMo Electronics Corporation,Taiwan)
Change from baseline of the percentage of vellus hair | Baseline (T0), 1 month (T1), 3 months (T3)
  Percentage of vellus hair (terminal hair has a diameter <0.04 mm) is calculate by Image-Pro Plus software on the microscopic images captured with Dino-Lite (AnMo Electronics Corporation,Taiwan)
Change from baseline of hair regrowth speed | Baseline (T0), 1 month (T1), 3 months (T3)
  Hair regrowth speed (mm/die) is calculate by Image-Pro Plus software on the microscopic images captured with Dino-Lite (AnMo Electronics Corporation,Taiwan)

SECONDARY OUTCOMES:
Change from baseline of superficial skin hydration | Baseline (T0), 1 month (T1), 3 months (T3)
  Skin electrical capacitance value is measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany).
  The measure of the skin capacitance properties is an indirect expression of its hydration level.

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy